CLINICAL TRIAL: NCT02685657
Title: A Phase II Randomized Multicenter Open Label Prospective Study of Neoadjuvant Chemotherapy Docetaxel With or Without MEK Inhibitor SELUMETINIB in Patients With Early and Locally Advanced Triple Negative Breast Cancer
Brief Title: Neoadjuvant Chemotherapy Docetaxel With or Without SELUMETINIB in Patients With Triple Negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Russian Academy of Medical Sciences (Other)
Collaborators: Russian Society of Clinical Oncology (Unknown)
Responsible Party: Principal Investigator, Mona Frolova, Senior Research Associate, Russian Cancer Research Center, Russian Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-14-10735
Record Dates: First submitted 2016-02-13; First posted 2016-02-19 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — AZD 6244; Doxorubicin; Cyclophosphamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AC followed by Docetaxel with Selumetinib (Experimental): Doxorubicin 60 mg/m2 and Cyclophosphamide 600 mg/m2 as a single IV infusion on day 1 of every 3 week cycle then 75 mg/m2 of Docetaxel given as a single IV infusion on day 1 of every 3 week cycle, 75 mg of SELUMETINIB twice a day PO on days 1-21 of every 3 week cycle
  Interventions: Drug: Drug: Selumetinib; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Docetaxel
- AC followed by Docetaxel (Active Comparator): Doxorubicin 60 mg/m2 and Cyclophosphamide 600 mg/m2 as a single IV infusion on day 1 of every 3 week cycle then 75 mg/m2 of Docetaxel given as a single IV infusion on day 1 of every 3 week cycle
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Docetaxel

INTERVENTIONS:
Drug: Drug: Selumetinib
  Other Names: AZD6244
  Arms: AC followed by Docetaxel with Selumetinib
Drug: Doxorubicin
Drug: Cyclophosphamide
Drug: Docetaxel

SUMMARY:
The purpose of this study is to increase survival of patients with early and locally advanced triple-negative breast cancer adding selumatinib to standard preoperative chemotherapy regimen.

DETAILED DESCRIPTION:
Molecular analysis of residual tumor after administration of neoadjuvant chemotherapy revealed several mechanisms of resistance to treatment. High frequency of RAS-RAF-MEK-ERK signal pathway activation was found in cells of triple negative breast cancer after neoadjuvant chemotherapy, which correlated with high proliferation index and low pathological complete response rate. Thus, inhibition of MEK molecule - an intermediary transducer of this pathway may decrease activity of this pathway and restore tumor sensitivity to cytostatic agents.

Hence, the use of SELUMETINIB, an oral selective inhibitor of MEK1/MEK2 kinases, in combination with Docetaxel should increase pathological complete response rate and in turn increase survival of patients with early and locally advanced triple-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* • Written informed consent;

  * Women with early and locally advanced breast cancer ( Stage IIB-IIIB: T2N1-2, T3-4/N0-2 or any T/N2)
  * Triple negative breast cancer (absence of estrogen receptor (0-2 points), progesterone receptor (0-2 points), and HER2/neu receptor (IHC 0-1+ or IHC 2+ in the absence of her2/neu gene amplification as evidenced by FISH);
  * Age: over 18 years;
  * Eastern Cooperative Oncology Group (ECOG) score: 0-1 points;
  * Left ventricular ejection fraction (LVEF) based on Echocardiogram (ECHO) or Multigated radionuclide angiography (MUGA scan): >55%
  * Laboratory values before the study start must meet the following criteria:

Absolute neutrophil count > 1500/microlitre Platelet count > 100000/microlitre Hemoglobin level > 9.0 g/dl Albumin > 2,5 g/dl Normal plasma creatinine level or estimated glomerular filtration rate (eGFR) >60 ml/minute Total bilirubin level < 1.25 upper limit of normal (ULN) Aspartate aminotransferase (AST), alanine aminotransferase (ALT) < 3 x ULN;

* Patient is able to abide by the protocol requirements (in the opinion of the Investigator)
* Patient's and her sexual partner's willing to use reliable methods of contraception (condoms with spermicidal foams/gels, intrauterine device) during the study and for at least 4 weeks after discontinuation of study treatment.
* Negative serum pregnancy test for women with childbearing potential or evidence of a post-menopausal status (total cessation of menses for more than 1 year. The following age-specific requirements must also apply:

  * Women < 60 years old: they would be considered post-menopausal if they have been amenorrheic for the past 12 months or more. The levels of Follicle-Stimulating Hormone (FSH) and estradiol must also be in the post-menopausal range (as per the institution).
  * Women ≥ 60 years;
  * Bilateral oophorectomy.

Exclusion Criteria:

* • Prior treatment (chemo-, hormone, radiation or immunotherapy) of breast cancer

  * Major surgery within 28 days prior to enrollment;
  * Known hypersensitivity to Docetaxel, SELUMETINIB or to the components of the investigational product;
  * Cardiac conditions as follows:

    a. Uncontrolled hypertension (BP ≥ 150/95 mmHg despite medical therapy) b. Acute coronary syndrome within 6 months prior to starting treatment c. Uncontrolled Angina - Canadian Cardiovascular Society grade II-IV despite medical therapy (Appendix 3) d. Symptomatic heart failure New York Heart Association (NYHA) Class II-IV, prior or current cardiomyopathy (Appendix 4) e. Prior or current cardiomyopathy including but not limited to the following: i. Known hypertrophic cardiomyopathy ii. Known arrhythmogenic right ventricular cardiomyopathy iii. Previous moderate or severe impairment of left ventricular systolic function (Left ventricular ejection fraction (LVEF) <45% on echocardiography or equivalent on MuGA) even if full recovery has occurred.

    f. Severe valvular heart disease g. Baseline Left ventricular ejection fraction (LVEF) below the lower limit of normal (LLN) or <55% measured by echocardiography or institution's LLN for MUGA h. Atrial fibrillation with a ventricular rate >100 bpm on ECG at rest i. QTcF >450ms or other factors that increase the risk of QT prolongation
  * Pregnancy or lactation;
  * Conditions (dementia, psychiatric or neurological disorders, drug addiction, alcoholism etc.) that limit patient's ability to undergo study procedures;
  * Simultaneous participation in other clinical studies;
  * Presence of acute or active chronic infections or other conditions (e.g. unstable or uncompensated respiratory, cardiac, hepatic, or renal disease, active bleeding diatheses or renal transplant), that in investigator's opinion may interfere with the treatment described in the study protocol;
  * Have refractory nausea and vomiting, chronic gastrointestinal diseases (e.g., inflammatory bowel disease), or significant bowel resection that would adversely affect the absorption / bioavailability of the orally administered study medication
  * History of another neoplasm (with the exception of adequately treated basal cell or cervical cancer in situ and cases when a cancer has been in remission for 5 years of more)
  * Ophthalmological conditions as follows:
* Intra-ocular pressure >21 mmHg, or uncontrolled glaucoma (irrespective of intra-ocular pressure)
* Current or past history of retinal pigment epithelial detachment / central serous retinopathy
* Current or past history of retinal vein occlusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
• Pathological complete response rate | After 24 weeks of neoadjuvant chemotherapy and surgery

SECONDARY OUTCOMES:
• Overall clinical response rate | After 24 weeks of neoadjuvant chemotherapy
• Adverse events rate in both treatment groups | After 24 weeks of neoadjuvant chemotherapy

OTHER OUTCOMES:
Association between RAS-ERK signal pathway activity in tumor and pathological complete response rate in patients who were receiving or not receiving SELUMETINIB | After 24 weeks of neoadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Mona Frolova, Principal Investigator — Russian Cancer Research Center

IPD SHARING:
Plan to Share IPD: No